CLINICAL TRIAL: NCT04045678
Title: A Randomized, Double-blinded, Multiple Ascending Dose Study in Patients With Early-stage Parkinson's Disease to Evaluate the Pharmacokinetics and Safety of LY03003 Following Intramuscular Injections
Brief Title: A Multiple Ascending Dose Study With LY03003 in Patients With Early-stage Parkinson's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Luye Pharma Group Ltd. (Industry)
Collaborators: Beijing Bozhiyin T&S Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LY03003/CT-CHN-103
Record Dates: First submitted 2019-07-30; First posted 2019-08-05 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Parkinson Disease
Keywords: parkinson disease; LY03003
MeSH Terms: conditions — Parkinson Disease | interventions — rotigotine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LY03003 (Experimental)
  Interventions: Drug: LY03003 ( Rotigotine, extended-release microspheres)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo, extended-release microspheres

INTERVENTIONS:
Drug: LY03003 ( Rotigotine, extended-release microspheres) — Patients to be enrolled to 70 mg dose group will receive 14 mg in the first week, 28 mg in the second week, 42 mg in the third week,56 mg in the fourth week and then 70 mg in the next 5 weeks.
  Patients to be enrolled to 84 mg dose group will receive 14 mg in the first week, 28 mg in the second week, 42 mg in the third week,56 mg in the fourth week, 70mg in the fifth week and then 84 mg in the next 5 weeks.
  Arms: LY03003
Drug: Placebo, extended-release microspheres — Patients to be enrolled to 70 mg dose group will receive 14 mg in the first week, 28 mg in the second week, 42 mg in the third week,56 mg in the fourth week and then 70 mg in the next 5 weeks.
  Patients to be enrolled to 84 mg dose group will receive 14 mg in the first week, 28 mg in the second week, 42 mg in the third week,56 mg in the fourth week, 70mg in the fifth week and then 84 mg in the next 5 weeks.
  Arms: Placebo

SUMMARY:
This study is to evaluate the safety and tolerability and to characterize the pharmacokinetics of multiple ascending dose (MAD) of LY03003 following intramuscular injections.

ELIGIBILITY:
Inclusion Criteria:

1. Patient had Parkinson's Disease that meet the clinical diagnostic criteria of the brain bank of the Parkinson's Disease Association of the United Kingdom.
2. Patient was Hoehn & Yahr stage ≤3 (excluding stage 0) ;
3. Patient was male or female aged 18 to 75 years;
4. Patient had a Mini Mental State Examination (MMSE) score of ≥25;
5. Patient had a Unified Parkinson's Disease Rating Scale (UPDRS) motor score (Part III) of ≥10 but ≤30 at Screening.
6. Patient who signed the informed consent form volunteered to participate in this clinical trial and could cooperate with the prescribed inspections.

Exclusion Criteria:

1. Patient had atypical Parkinson's syndrome(s) due to drugs (e.g., metoclopramide, flunarizine), metabolic neurogenetic disorders (e.g., Wilson's disease), encephalitis, cerebrovascular disease, or degenerative disease (e.g., progressive supranuclear palsy);
2. Patient had a history of pallidotomy, thalamotomy, deep brain stimulation, or fetal tissue transplant;
3. Patient had dementia, schizophrenia or hallucinations, or clinically significant depression;
4. Patient had a lifetime history of suicide attempt (including an active attempt, interrupted attempt, or aborted attempt), or presence of suicidal ideation in the past 6 months as indicated by a positive response ("Yes") to either Question 4 or Question 5 of the Columbia-Suicide Severity Rating Scale (C-SSRS) at Screening;
5. Patient had a history of orthostatic hypotension with a decrease of ≥20 mmHg in systolic blood pressure (SBP) or ≥10 mmHg in diastolic blood pressure when changing from the supine to the standing position and keeping in the standing position for 3 minutes;
6. Patient had received therapy with a dopamine (DA) agonist either concurrently or had done so within 28 days prior to the Screening;
7. Patient had received therapy with 1 of the following drugs either concurrently or within 28 days prior to Screening: monoamine oxidase B (MAO-B) inhibitors (e.g., pargyline, selegiline), DA releasing agents (e.g., amphetamine), reserpine, DA-antagonists (e.g., metoclopramide), neuroleptics, or other medications that may interact with DA function;
8. Patient was currently (at the time of Screening) receiving central nervous system active therapy (e.g., sedatives, hypnotics, antidepressants, anxiolytics), unless the dose had been stable for at least 28 days prior to Screening Visit and was likely to remain stable for the duration of the study;
9. Patient had a current diagnosis of epilepsy, had a history of seizures as an adult within 1 year prior to Screening, had a history of stroke or transient ischemic attack within 3 months prior to Screening;
10. Patient had a history of known intolerance/hypersensitivity to non-dopaminergic antiemetics, such as domperidone, ondansetron, tropisetron;
11. Patient had clinically significant liver dysfunction (which defined as total bilirubin above the upper limit of normal range, or alanine transferase (ALT) and / or aspartate transferase (AST) 2 times higher than the upper limit of normal range);
12. Patient had clinically significant renal insufficiency (serum creatinine >2.0 mg/dL [ >178 μmol/L]);
13. Patient had clinically significant cardiac insufficiency and/or had myocardial infarction in the past 12 months;
14. Patient had a history of allergic to any medication;
15. Heavy smoker, alcoholic, drug addict;
16. Female patients who were pregnant or were breastfeeding or were of childbearing potential without adequate contraception; male patients who cannot take adequate contraception during the study;
17. Patient who was inappropriate to participant in the study in the judgment of the Investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-10-10 (Actual); Primary Completion 2019-04-16 (Actual); Study Completion 2019-06-21 (Actual)

PRIMARY OUTCOMES:
Frequency of adverse events | From screening up to day 50
  Adverse events to evaluate the safety and tolerability of LY03003

SECONDARY OUTCOMES:
Time of maximum concentration (Tmax) of total LY03003 | From the first injection of stable doses up to day 50
Maximum concentration in plasma (Cmax) of total LY03003 | From the first injection of stable doses up to day 50
Area under the concentration-time curve (AUC) from zero up to the last measured concentration [AUC (0-t)] of LY03003 | From the first injection of stable doses up to day 50
Area under the concentration-time curve (AUC) from time zero up to the infinite time [AUC (0-∞)] of LY03003 | From the first injection of stable doses up to day 50
Apparent volume of distribution (Vd) of LY03003 | From the first injection of stable doses up to day 50
Terminal half-life (t1/2) of total LY03003 | From the first injection of stable doses up to day 50
Total body clearance of LY03003 | From the first injection of stable doses up to day 50
Maximum steady-state drug concentration of LY03003 | From the first injection of stable doses up to day 50
Minimum steady-state drug concentration of LY03003 | From the first injection of stable doses up to day 50
Average steady-state concentration of LY03003 | From the first injection of stable doses up to day 50
Area under the concentration-time curve (AUC) at steady-state concentration of LY03003 | From the first injection of stable doses up to day 50
Fluctuation degree in steady-state concentration of LY03003 | From the first injection of stable doses up to day 50
Change from baseline to the end of the treatment period in the Unified Parkinson's Disease Rating Scale (UPDRS) part (Ⅱ+Ⅲ) Total Score | Screening, baseline, days 29 and day 50
  The Unified Parkinson´s Disease Rating Scale Part Ⅱ measures "Activities in Daily Living". The total score ranges from 0 (Best score possible) to 52 (Worst score possible).
  The Unified Parkinson´s Disease Rating Scale Part Ⅲ is an accepted and validated scale for the assessment of motor function in Parkinson´s disease. Each of the 27 sub-items in the UPDRS III is measured on a scale of 0 to 4, where 0 is normal and 4 represents severe abnormalities. The total scores therefore ranges from 0 to 108.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Chinese PLA General Hospital, Beijing
  - Xuanwu Hospital Capital Medical University, Beijing
  - Shengjing Hospital of China Medical University, Shenyang